CLINICAL TRIAL: NCT03413982
Title: Bladder Cancer Longitudinal Biorepository for Development of Novel Therapeutics/Biomarkers
Acronym: GUB-BCR-001
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00141546
Record Dates: First submitted 2018-01-10; First posted 2018-01-29 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples Without DNA — Blood, urine, and tissue are being collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BC Patients: Patients with bladder cancer. This registry involves no intervention. Blood, urine, and tissue samples will be collected to be used for research.
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry — Patient registry

SUMMARY:
The purpose of this study is to create a registry, which is a "bank" of information about patients who have had similar medical conditions and treatments. The registry will be used by researchers to learn more about long term outcome of patients with bladder cancer, how bladder cancer tissues are related to tumor development, recurrence and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to clinic with presumed bladder cancer or have a diagnosis of bladder cancer are eligible to participate
* Patients can participate in any additional research studies during the patients' participation within this protocol.

Exclusion Criteria:

* Patients who do not have presumed bladder cancer will not be eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are receiving care from KUMC clinics will be considered for this registry.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-11-02 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Blood, urine and tissue characteristics of bladder cancer patients | 24 months
  Samples will be collected over a 24 month period for patients to build a biorepository for future research on how they are related to tumor development, recurrence and survival.

CONTACTS AND LOCATIONS:
Overall Officials: John Taylor, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States